CLINICAL TRIAL: NCT05756556
Title: A Phase 2a, Open-label Study of T3011 in Combination With Cobimetinib in Patients With Advanced Melanoma
Brief Title: T3011 in Combination With Cobimetinib in Patients With Advanced Melanoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in drug development and lifecycle management and decide to suspend this study
Sponsor: ImmVira Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVR-T3011-IT-2004
Record Dates: First submitted 2022-12-23; First posted 2023-03-06 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Melanoma; Malignant Melanoma
Keywords: intratumoral (IT) injection; Cobimetinib; advanced melanoma; RAS mutation-positive; BRAF V600E/V600K mutation-positive; stage IIIB to IV advanced malignant melanoma
MeSH Terms: conditions — Melanoma | interventions — cobimetinib

STUDY DESIGN:
Intervention Model Description: This is a phase 2a, open-label study of T3011 given via intratumoral (IT) injection in combination with Cobimetinib given via oral administration in patients with advanced melanoma. This study is planned to enroll approximately 62~68 patients with BRAF V600E/V600K mutation-positive or RAS mutation-positive, which will be conducted in 2 parts (part 1 and part 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 2a (Experimental): T3011 given via intratumoral (IT) injection in combination with Cobimetinib via oral administration in patients with advanced melanoma.
  Interventions: Combination Product: T3011 + Cobimetinib

INTERVENTIONS:
Combination Product: T3011 + Cobimetinib — 1e8 plaque-forming units (PFU)/mL (up to 10 mL, every 2 weeks [Q2W], 28 days/cycle) T3011 will be administered in combination with 60 mg Cobimetinib (once daily [QD] for the first 21 days of each 28-day cycle)

SUMMARY:
This study will evaluate the efficacy and safety of T3011 in combination with Cobimetinib in patients with advanced melanoma.

DETAILED DESCRIPTION:
This is a phase 2a, open-label study of T3011 given via intratumoral (IT) injection in combination with Cobimetinib given via oral administration in patients with advanced melanoma. This study is planned to enroll approximately 62~68 patients with BRAF V600E/V600K mutation-positive or RAS mutation-positive, which will be conducted in 2 parts (part 1 and part 2).

ELIGIBILITY:
Inclusion Criteria

All patients must meet the following criteria for inclusion:

1. Patient has provided informed consent prior to initiation of any study-specific activities/procedures.
2. Male or female age ≥ 18 years at the time of informed consent.
3. Willingness to provide pre-and post-treatment fresh tumor biopsy specimens as specified in the Schedule of Study Procedures and Assessments (Table 1).
4. Histologically confirmed diagnosis of malignant melanoma (except for uveal melanoma).
5. Patient with stage IIIB to IV advanced malignant melanoma (as defined by American Joint Committee on Cancer [AJCC] staging manual version 8.0) that is not surgically resectable, failed for standard of care (SOC) therapy or in the opinion of the investigator not suitable for SOC therapy. SOC may include, but not be limited to chemotherapy, targeted therapy or immunotherapy.
6. BRAF V600E/V600K mutation-positive (applied to part 1 and part 2 cohort 1) or RAS mutation-positive (applied to part 1 and part 2 cohort 2). BRAF V600E/V600K and RAS mutation status result from diagnosis of tumor histopathology should be provided during Screening. If the patient is unable to provide, testing will be required during the Screening period in local laboratory.
7. Measurable disease defined as one or both of the following:

（1） At least 1 melanoma lesion that can be accurately and serially measured in at least 2 dimensions sand for which the longest diameter is ≥ 10 mm and with perpendicular diameter ≥ 5 mm as measured by contrast-enhanced or spiral CT scan for visceral or nodal/soft tissue disease. Lymph nodes must measure > 15 mm in their short axis to be considered measurable by CT scan.

（2） At least 1 superficial cutaneous or subcutaneous melanoma lesion that can be accurately and serially measured in at least 2 dimensions and for which the short axis is ≥ 5 mm as measured by calipers.

（3） Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that lesion since radiation.

8. Injectable disease (i.e., suitable for direct injection or through the use of ultrasound [US] or CT guidance) defined as follows:

1. At least 1 injectable melanoma lesion ≥ 5 mm in longest diameter, or in the opinion of the investigator the lesion can be injected.

9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

10. Life expectancy ≥ 12 weeks.

11. Adequate bone marrow function defined by ANC of ≥ 1.5 × 109/L, platelet count of ≥ 100 × 109/L, and hemoglobin (Hb) of ≥ 8.5 g/dL.

12. Adequate hepatic function defined as AST/ALT ≤ 3 × ULN and total bilirubin ≤ 1.5 × ULN (except patients with Gilbert's Syndrome, wherein total bilirubin < 3.0 mg/dL is acceptable; patients with hepatic metastases: AST and/or ALT ≥ 5 × ULN is acceptable; patients with hepatic or bone metastases: ALP ≥ 5 × ULN is acceptable).

13. Adequate renal function defined as creatinine clearance > 50 mL/min as determined by the Cockcroft-Gault equation.

14. Adequate coagulation function defined as international normalization ratio (INR)/prothrombin time (PT) ≤ 1.5 × ULN, and partial thromboplastin time (PTT)/ activated PTT (aPTT) ≤ 1.5 × ULN, unless the patient is receiving anticoagulant therapy, in which case PT and PTT/aPTT must be within therapeutic range of intended use of anticoagulants.

15. Resolution of all prior anti-tumor therapy toxicities (except for alopecia) to ≤ NCI CTCAE version 5.0 Grade 1.

Note: patients with immune-mediated endocrinopathies on replacement therapy are eligible. Patients with endocrine-related AE who can recover to ≤ NCI CTCAE version 5.0 Grade 1 after hormone replacement therapy, in the judgment of the investigator, have no impact on the safety and efficacy of this study can also be enrolled. Patients with toxicities attributed to the prior anti-tumor therapy and not expected to resolve, such as neuropathy or ototoxicity after platinum-based therapy, are permitted to enroll. Patients with other toxicities > NCI CTCAE version 5.0 Grade 1 may be enrolled with approval from the sponsor.

16. Female patients must be surgically sterile (or have a monogamous partner who is surgically sterile), or be at least 2 years postmenopausal, or commit to using 2 acceptable forms of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives, or abstinence) for the duration of the study and for 6 months following the last dose of study treatment. Male patients must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study and for 6 months following the last dose of study treatment.

17. Women of childbearing potential (WCBP) must have a negative serum pregnancy test at Screening within 14 days before the first dose of study treatment on W1D1 and a negative urine pregnancy test pre-dose on W1D1 (assessment not required at W1D1 if completed within the previous 7 days of W1D1).

Note: A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis).

Exclusion Criteria

Patients are to be excluded from the study if they meet any of the following criteria:

1. Prior treatment with other Oncolytic virus (OV) (including but not be limited to T-VEC), tumor vaccines, cellular therapy or gene therapy.
2. Prior local anti-tumor therapy < 21 days prior to the first dose of study treatment; prior systemic targeted therapy (including but not be limited to MEK inhibitors) < 21 days or last dose of therapy with MEK inhibitors < 5 times the half-life prior to first dose of study treatment; prior other anti-tumor therapy (including but not be limited to PD-1/programmed cell death ligand 1[PD-L1]) < 21 days prior to the first dose of study treatment, prior major surgery < 21 days prior to the first dose of study treatment.
3. Prior treatment with anti-PD-(L)1 monoclonal Ab in combination with IL-12.
4. Previous intolerance to anti-PD-(L)1 monoclonal Ab or previous history of immunotherapy induced ≥ NCI CTCAE version 5.0 Grade 3 non-infectious pneumonitis/interstitial lung disease.
5. The following foods/supplements are used within 7 days before the study treatment or the following foods/supplements are planned to be used during the study treatment:

（1） St. John's wort or hyperforin (potent cytochrome P450 CYP3A4 enzyme inducer).

（2） Grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor).

6. Refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection that would interfere with absorption of study drugs, inability or unwillingness to swallow the formulated product.

7. A history of metastasis to the brain stem, midbrain, pons/medulla oblongata, or within 10 mm of optic nerve organs (optic nerve and optic chiasma); Or a history of leptomeningeal metastasis.

8. Patients with rapidly disease progression, defined as patients who cannot tolerate interruption of systemic anti-tumor therapy for at least 8 weeks, according to the investigator's judgment.

9. Primary or acquired immunodeficient status (leukemia, lymphoma, human immunodeficiency virus [HIV]/acquired immunodeficiency syndrome [AIDS]).

10. History or evidence of active autoimmune disease that requires systemic treatment (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs) within 4 weeks prior to first dose of study treatment. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

11. History or evidence of active primary immunodeficiency. 12. Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug. The following are exceptions to this criterion:

1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection).
2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).

13. Requires continued concurrent systemic therapy with any drug active against herpes simplex virus (HSV) (acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir). Topical use of drugs against HSV are allowed.

14. Live, attenuated vaccines within 4 weeks prior to initiation of study treatment (patients vaccinated with inactivated vaccines can be enrolled).

15. Active infection requiring systemic treatment. 16. Hepatic diseases known to be clinically significant include alcoholism, cirrhosis, fatty hepatic disease, and other hereditary hepatic diseases, or positive serological test of hepatitis B virus (HBV) or hepatitis C virus (HCV) at Screening.

1. Patients who test positive for anti-hepatitis C Ab (anti-HCV) but negative for HCV ribonucleic acid (RNA) are considered eligible to participate in the study.
2. Patients with infection of hepatitis B (positive hepatitis B surface antigen [HBsAg] result) will be excluded. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core Ab [HBcAb] and absence of HBsAg) are eligible.

17. Female patient is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 6 months after the last dose of study treatment.

18. History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, central serous chorioretinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration. Patients will be excluded from study participation if they currently are known to have any of the following risk factors for RVO:

1. History of serous retinopathy;
2. History of retinal vein occlusion;
3. Evidence of ongoing serous retinopathy or RVO at baseline.

19. Patients with active central nervous system (CNS) lesions (i.e., those with radiographically unstable, symptomatic lesions, including but not limited to carcinomatous meningitis) and history of intracranial hemorrhage are excluded. However, patients are eligible if:

1. Patients with all known CNS lesions have been treated with stereotactic therapy or surgery, whose disease is stable without using corticosteroids; AND
2. There has been no evidence of clinical and radiographic disease progression in the CNS for ≥ 3 weeks after radiotherapy or surgery.

20. History of another primary malignant tumor, except the following: 1) the patient has undergone potentially curative therapy with no evidence of that disease and recurrence for 3 years prior to the first dose of study treatment; 2) Adequately treated non-melanoma skin cancer or lentigo with no evidence of malignancy; 3) Adequately treated carcinoma in situ without evidence of disease.

21. Patients with moderate to large amount of pleural effusion, ascites or pericardial effusion who need drug or medical intervention. Patient may be eligible to participate following discussion with investigator and approval from the sponsor.

22. Unexplained > 38.5℃ fever (If the fever is caused by the tumor according to the investigator's judgment, the patient can be enrolled) occurs during the Screening period or on the day of administration, which in the judgment of investigator, would interfere with patient participation in the study or evaluation of patient's efficacy.

23. History of seizure disorders within 6 months prior to Screening. 24. Active oral or skin herpes lesion at Screening. 25. Plan to receive any other anti-tumor therapy (including herbal therapy that has anti-tumor effects) during treatment with study drug.

26. History of congestive heart failure (> New York Heart Association Class II), active coronary artery disease, unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest), LVEF below institutional lower limit of normal or below 50%, whichever is lower, poorly controlled hypertension, defined as sustained, uncontrolled, nonepisodic baseline hypertension consistently above 159/99 mmHg despite optimal medical management, or clinically significant cardiac arrhythmias.

27. Uncontrolled diabetes or symptomatic hyperglycemia. 28. History of allergic reactions attributed to compounds of similar biological composition to HSV-1, IL-12, or anti-PD-1 monoclonal Ab or their excipients.

29. History of psychiatric disorders that would interfere with cooperation with the requirements of the trial or is still requiring for medication control.

30. History of substance abuse (including alcohol) within 6 months prior to signing informed consent.

31. Other systemic conditions or organ abnormalities that, in the opinion of the investigator, may interfere with the conduct and/or interpretation of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 5 years after the first dose of the last patient, depending on the actual situation.
  defined as the proportion of patients with a CR or PR on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to RECIST version 1.1
Characterize the safety and tolerability of T3011 in combination with Cobimetinib. | up to 5 years after the first dose of the last patient, depending on the actual situation.
  Incidence and severity of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), dose-limiting toxicities (DLTs) (part 1 only), adverse event of special interest (AESIs), abnormal clinically significant vital signs, physical examination, and laboratory tests, with severity determined according to national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 5 years after the first dose of the last patient, depending on the actual situation.
  defined as the time from initiation of study treatment to death from any cause
Progression-free survival (PFS) | up to 5 years after the first dose of the last patient, depending on the actual situation.
  defined as the time from initiation of study treatment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST version 1.1
Disease control rate (DCR) | up to 5 years after the first dose of the last patient, depending on the actual situation.
  defined as the proportion of patients who have a best overall response of CR or PR or SD, as determined by the investigator according to RECIST version 1.1.
Duration of response (DOR) | up to 5 years after the first dose of the last patient, depending on the actual situation.
  defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST version 1.1.
European Organization for Research and Treatment of Cancer Questionnaire Core 30 (EORTC QLQ-C30) | up to 5 years after the first dose of the last patient, depending on the actual situation.
  Change from baseline in the European Organization for Research and Treatment of Cancer Questionnaire Core 30 (EORTC QLQ-C30) (version 3.0) at subsequent visits protocol required.

CONTACTS AND LOCATIONS:
Locations (1):
- Gabrail Cancer and Research Center, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No